CLINICAL TRIAL: NCT04548687
Title: Pilot Prospective Randomized Clinical Trial "Insufflation of Carbon Dioxide During Minimally Invasive and Repeated Cardiac Surgery"
Brief Title: a Randomized Clinical Trial Evaluating the Effectiveness of Carbon Dioxide Use in Cardiac Surgery
Acronym: CAR-DRIVER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 496
Record Dates: First submitted 2020-09-01; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-06

CONDITIONS: Carbon Dioxide
Keywords: carbon dioxide; cardiac surgery; delirium; minimally invasive intervention; redo cardiac surgery
MeSH Terms: conditions — Delirium | interventions — Carbon Dioxide

STUDY DESIGN:
Intervention Model Description: Group 1: patients with planned minimally invasive or repeated cardiac surgery using standard methods of deaeration of cardiac cavities.
  Group 2: patients with planned minimally invasive or repeated cardiac surgery using standard methods of deaeration of cardiac cavities, supplemented with carbon dioxide insufflation during surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- carbon dioxide insufflation (Active Comparator): patients with planned minimally invasive or repeated cardiac surgery using standard methods of deaeration of cardiac cavities, supplemented with carbon dioxide insufflation during surgery + standard methods of deaeration of cardiac cavities
  Interventions: Procedure: carbon dioxide insufflation
- no carbon dioxide (Other): standard methods of deaeration of cardiac cavities: manual method, change in body position, through the cannula of the ascending aorta, through the drainage of the left ventricle
  Interventions: Procedure: No carbon dioxide insufflation

INTERVENTIONS:
Procedure: carbon dioxide insufflation — Carbon dioxide insufflation at a rate of 5 l / min. through the Redon drainage during cardiac surgery (minimally invasive or repeated) during cardiopulmonary bypass
  Other Names: carbon dioxide
  Arms: carbon dioxide insufflation
Procedure: No carbon dioxide insufflation — standard methods of deaeration of cardiac cavities: manual method, change in body position, through the cannula of the ascending aorta, through the drainage of the left ventricle
  Other Names: standard methods of deaeration
  Arms: no carbon dioxide

SUMMARY:
study of the efficacy and safety of carbon dioxide in cardiac surgery: repeated or minimally invasive

DETAILED DESCRIPTION:
prospective randomized clinical single-center study of the efficacy and safety of using carbon dioxide in deaeration of cardiac cavities during cardiac surgery (repeated interventions and minimally invasive interventions)

ELIGIBILITY:
Inclusion Criteria:

* Planned cardiac surgery on the left heart with limited deaeration: Minimally invasive approach (mininotomy, minimally invasive lateral thoracotomy); Re-intervention
* Signed informed voluntary consent

Exclusion Criteria:

* Patient refusal to participate in any stage of the study
* History of stroke, transient ischemic attack
* Hemodynamically significant stenosis of the brachiocephalic arteries (more than 70%)
* Swelling or thrombosis of the heart
* LV dysfunction (EF less than 30%)
* Atherosclerosis of the aorta (atheromatosis)
* Surgical access conversion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-06-20 (Estimated); Study Completion 2022-06-20 (Estimated)

PRIMARY OUTCOMES:
delirium: CAM-ICU, 3-D CAM | 7 days after surgery
  positive test development of postoperative delirium: Richmond Agitation-Sedation Scale, Confusion Assessment Method-Intensive Care Unit (more than one error) - while in the intensive care unit; positive test the 3-Minute Diagnostic Interview for Confusion Assessment Method (CAM) defined delirium - while in the ward of the department: The CAM algorithm is considered positive if the following features are present: Feature 1) Acute onset or fluctuating course and Feature 2) Inattention and either Feature 3) Disorganized thinking or Feature 4) Altered level of consciousness.

SECONDARY OUTCOMES:
deaeration time | intraoperatively
  deaeration time according to transesophageal echocardiography data
neurocognitive dysfunction | 7 days after surgery
  development of neurocognitive dysfunction: Montreal Cognitive Assessment - two days before surgery and 7 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexander V. Bogachev-Prokophiev, MD, PhD, Principal Investigator — E.Meshalkin National medical research center
Locations (1):
- "E.Meshalkin National medical research center" of the Ministry of Health of the Russian Federation, Novosibirsk, Russia